CLINICAL TRIAL: NCT03850262
Title: Role of MRI in Traumatic Posterolateral Corner Of The Knee
Brief Title: Traumatic Posterolateral Corner Of The Knee
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alice Mansour Louis, principal investigator, Assiut University
Other Study IDs: Traumatic knee
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Traumatic Posterolateral Corner Of The Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with posterolateral corner trauma of the knee
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — The study will be done on 1.5T MR unit (Siemens) and 1.5T MR unit (Philips) at Assuit University Hospital, or 1.5T MR unit (G.E.) at Eman General Hospital.
  * The field of view varied between 14 cm and 16 cm, and slice thickness varied between 3 and 4 mm, with 0.5 mm intersection gap.
  * Imaging sequences included sagittal PD proton density, T2 and STIR, axial PD, coronal STIR and coronal oblique.

SUMMARY:
The posterolateral corner (PLC) is known as the "dark side of the knee" due to its complex and variable anatomy.Its stability is provided by capsular and non-capsular structures that function as static and dynamic stabilizers.

The structures of the PLC are primarily responsible for resisting varus angulation and external tibial rotation. They also act as secondary stabilizers, in conjunction with the cruciate ligaments, to prevent anterior and posterior translation during the early phase of flexion (0°-30°) PLC injures are relatively uncommon, occurring in approximately 16% of all knee injuries. They are rarely seen in isolation, as the majority is associated with concomitant cruciate ligament tears, as well as meniscal tears and injuries to the medial ligamentous structure.

DETAILED DESCRIPTION:
The mechanism of injuries is commonly result of a posterolaterally directed blow to the anteromedial aspect of the proximal tibia with the knee in full extension, other less common mechanisms include posterior rotatory dislocation (dashboard injury), anterior rotatory dislocation, and hyperextension injury with external rotation.

Early diagnosis of injuries to the posterolateral aspect of the knee is critical because surgical repair in the acute period is easier, and is associated with a more favorable outcome for patients. Also, failure to address instability of the PLC structures increases forces at anterior cruciate ligament (ACL) and posterior cruciate ligament (PCL) graft sites and may lead to failure of the cruciate reconstruction ,significant osteoarthritis and chronic knee instability Since introduction of MRI to musculoskeletal imaging in the early 1980s, it has proven to be an excellent technique for evaluating patients with knee problems. Its main advantages of MRI are its non-invasive nature and its high accuracy and negative predictive value in evaluating the menisci and ACL. Also it is useful in the detection and diagnosis of various traumatic, non traumatic knee abnormalities and diagnosis of occult or unsuspected bone lesions. It can help in the selection of those patients who need therapeutic arthroscopy.

Assessment of PLC injures is usually made clinically , including several physical examination maneuvers by orthopedic physician ; such as posterolateral drawer test, dial test, reverse pivot shift test, external rotation recurvatum test and varus stress test.

Despite these several tests, in 72% of cases they are not identified in his initial presentation, which demonstrates the difficulty of clinical diagnosis.

Thus, it is important to use additional tests for the diagnosis of posterolateral corner injury. The medical literature demonstrates that MRI has an accuracy of up to 95% for identifying major injury PLC structures, namely, lesions of the lateral collateral ligament (LCL), popliteus muscle tendon (PMT) and poplitealfibular ligament (PFL).

For better visualization of the PLC structures, an oblique coronal T2 cut should be performed. It provides an accurate and detailed evaluation of the posterolateral corner structures of the knee.

As PLC injures may be difficult to be assessed clinically because of associated and coexisting injuries at the knee, so MRI can provide vital information regarding the status of the posterolateral corner, thus enabling good surgical planning and more effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have positive tests of posterolateral corner instability by clinical examination.
2. Patients who suspected by Plain X-ray to have posterolateral corner injury.

Exclusion Criteria:

1. Patients whom previously underwent arthroscopy or surgically intervention to knee joint.
2. Patients with history of fracture repaired by metal plates or screws.
3. Patients have phobia of indoor places.
4. Patients with contraindication to MRI like intra-cerebral aneurysmal clips, cardiac pacemaker, and metallic foreign body at region of examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with posterolateral corner trauma of the knee
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MRI in diagnosis of forty patients with posterolateral corner trauma of the knee. | one year
  MRI at Radiological department will be done to evaluate injuries of PLC posterolateral corner of the knee in correlation with clinical or operative findings (either open or arthroscopic) as gold standard.

REFERENCES:
- [Background] Fornalski S, McGarry MH, Csintalan RP, Fithian DC, Lee TQ. Biomechanical and anatomical assessment after knee hyperextension injury. Am J Sports Med. 2008 Jan;36(1):80-4. doi: 10.1177/0363546507308189. Epub 2007 Oct 11. PMID 17932409
- [Background] Baker CL Jr, Norwood LA, Hughston JC. Acute posterolateral rotatory instability of the knee. J Bone Joint Surg Am. 1983 Jun;65(5):614-8. PMID 6853566